CLINICAL TRIAL: NCT03499938
Title: Structured Light Plethysmography in Children Admitted Due to Acute Obstructive Airways Disease
Brief Title: Structured Light Plethysmography in Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Pneumacare Ltd (Industry); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 237151
Record Dates: First submitted 2018-03-26; First posted 2018-04-17 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pediatric Respiratory Diseases
Keywords: Asthma; Bronchiolitis; Wheezing; Structured Light Plethysmography
MeSH Terms: conditions — Asthma; Bronchiolitis; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Structured Light Plethysmography — Non-invasive non-contact measurement of tidal breathing during hospital admission

SUMMARY:
Obstructive airways disease is the most common group of acute illnesses leading to hospital treatment in children. This group consists of different age-related diagnoses, such as bronchiolitis in infants or wheezing and asthma in older children. Though these entities overlap with each other, they have common characteristics and the same leading symptom breathing distress.

The investigators aim conduct an observational cohort study to examine if the clinical course of respiratory distress be quantified and the treatment improved in children with acute breathing difficulty using a new non-touch non-invasive SLP measurement device?

Thora3Di is a new CE- and FDA-approved medical device able to measure chest and abdominal wall movements during tidal breathing with a method called structured light plethysmography (SLP). The method is non-touch and non- invasive, it does not need any connection with the child.

One-month- to 12-years-old infants and children are recruited from the paediatric wards at Evelina London Children's hospital. The child lies or sits within the field of vision of the SLP device with their chest and abdomen exposed. A grid pattern of normal light will be projected onto the chest and changes in the format of the grid as the infant or child breathes will be recorded by the SLP device. Data will be collected for each child for 3-5 minutes once in 24 hour periods for 2-10 times during hospital stay.

The aim is to reduce duration of hospital stay by finding predicting parameters for obstructive airways diseases with the new SLP method, and further aim to standardization of treatment strategies, to reduce expenditure.

DETAILED DESCRIPTION:
Cohort pilot study to characterise the chest wall movement during tidal breathing in children admitted due to acute obstructive airways disease, using non-invasive SLP methodology (Thora3DiTM).

The investigators propose to utilise the SLP in children admitted for obstructive airways disease and track progression of their condition during the hospital stay. Focus will be in the SLP output, and investigators aim to 1) quantify the breathing distress and whether this number has an effect on the patient outcome and 2) further aim to see if regional changes in the thoracic-abdominal movement can be recognized by the measurement method.

The data collected from this study will allow investigators to characterise chest wall movements in children with obstructive airways disease and to examine the effect of the treatment on this movement.

Study population

Investigators will aim to recruit:

* 35-60 children between the ages of 1 month and 12 years with acute obstructive airways disease
* Admitted to hospital within 24 hours

Locations: Participants are children, in Evelina Children's hospital as a patient due to obstructive airways disease

The eligible children admitted to hospital will be identified at the clinical handovers and after obtaining the parental consent to participate in the study, the first measurements are performed as soon as possible, however within the first 24 hours of admission. The SLP measurements are repeated in 24 hour intervals 2-10 times depending on the duration of hospital stay.

Clinical patient data of age, sex, ethnicity, weight and length will be collected. A member of the clinical / research team (respiratory clinical fellow) collects structured data on the breathing distress using a modified pulmonary index scale for children (mPIS).

Measurement of standard clinical variables, such as respiratory rate, heart rate and oxygen saturation will be made each time the SLP readings are recorded. The measurement will be taken on a bare skin with a white medical adhesive tape to cover any existing medical attachments on thoracic-abdominal region (such as ECG electrodes). Alternatively, measurements can be made if the child is wearing a close fitting white garment without any creases (such as a babygrow).

A structured light pattern will be projected onto the chest and abdominal wall and the movement of this pattern as the patient breathes will be recorded for 3-5 min. The total period of testing per session should take approximately 15 minutes per person, including the movement of the device and the positioning of the patient.

Physiological and clinical data collection at each study point:

Dates of onset of breathing difficulty, admission and discharge Oxygen treatment and breathing support (Flow in L/min for HFNC, Fi02 %O2, CPAP settings) Current medication Need for NG-tube Need for IV-fluids Heart Rate SaO2 Respiratory Rate

Data analysis will include the traditional time indices from tidal breathing, and the variability of these time indices.

Appropriate statistical analyses will be identified depending on the study and distribution of the samples (parametric vs. non-parametric). It is suspected that t-tests (one-sample to two sample), analysis of variance (ANOVA), or Mann-Whitney-U tests will be used where appropriate.

The investigators will also explore novel higher levels of data interpretation including Bayesian interpretation of respiratory function, and machine learning to predict disease diagnosis, severity and discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month to 12 years
* Any children who have been admitted to ELCH with a diagnosis of acute obstructive airways disease within 24 hours
* Weight over 3 kg

Exclusion Criteria:

* Weight less than 3kg
* History of thoracic or abdominal surgery, or any acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to participate in the study
* Patients with significant co-morbidities resulting in clinical instability (assessed by the clinician at screening only), such as diaphramatic dysfunction, tracheostomy or need for non-invasive or invasive ventilation

Ages: 1 Month to 12 Years | Sex: All
Age Groups: Child
Study Population: Children admitted to paediatric HDU/ICU wards for acute obstructive airways disease aged 1 month to 12 years
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Clinical severity of breathing distress measured by modified pulmonary index score (mPIS) | Change in clinical severity score during hospital admission. Data will be collected for each child once in 24 hour periods for 2-10 times during hospital stay.
  To examine whether SLP can predict clinical severity, the relationship between SLP tidal breathing parameters and clinical score (mPIS is a composite score from RR, HR, Sat02, Wheezing, Accessory muscle use, Inhalation-Exhalation-ratio) will be assessed. For each of these 6 measurements or observations, a score of 0 to 3 is assigned, resulting in a possible minimum score of 0 and a maximum score of 18. A cut-off score of 12 has been studied to distinguish more severe asthmatic exacerbation in children. (Carrol et al 2005) Primary outcome measure: mPIS

SECONDARY OUTCOMES:
Regional SLP tidal breathing parameters (relative contribution) | Change in SLP relative contribution during hospital admission. Data will be collected for each child once in 24 hour periods for 2-10 times during hospital stay.
  To characterise regional thoraco-abdominal movements in children with obstructive airways disease and to examine the effect of standard treatment procedures on this movement. Primary Outcome measure: Regional SLP tidal breathing parameter (relative contribution)
Regional SLP tidal breathing parameters (phase) | Change in SLP phase during hospital admission. Data will be collected for each child once in 24 hour periods for 2-10 times during hospital stay.
  To characterise regional thoraco-abdominal movements in children with obstructive airways disease and to examine the effect of standard treatment procedures on this movement. Primary Outcome measure: Regional SLP tidal breathing parameter (phase).

OTHER OUTCOMES:
Clinical outcome (Length of stay) | Length of stay is calculated as time from hospital admission (entering the primary ward) to time of hospital discharge (leaving the final ward). The estimated length of hospital stay will be a minimum of 1 and maximum of 30 days.
  To examine whether tidal breathing patterns can predict clinical outcome, the relationship between SLP tidal breathing parameters and clinical outcome (as measured by length of hospital stay [LOS]) will be assessed. Primary outcome measures: LOS

CONTACTS AND LOCATIONS:
Overall Officials: Richard Iles, Dr, Study Director — Guy´s and St Thomas´ NHS trust; Eero Lauhkonen, Dr, Principal Investigator — Guy´s and St Thomas´ NHS trust
Locations (1):
- Evelina London Children´s Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: P88 Structured light plethysmography in toddlers admitted due to acute wheezing — https://thorax.bmj.com/content/73/Suppl_4/A150.1
- See also: Using Adaptive Principal Component Analysis (APCA) and Machine Learning to characterise paediatric asthma in data collected by Structured Light Plethysmography (SLP) | European Respiratory Society — https://erj.ersjournals.com/content/54/suppl_63/PA922